CLINICAL TRIAL: NCT06262126
Title: A Feasibility Study of Virtual Reality for the Treatment of Non-cardiac Chest Pain
Brief Title: Virtual Reality for Non-cardiac Chest Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andree H. Koop, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-012673
Record Dates: First submitted 2024-01-25; First posted 2024-02-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Diseases; Chest Pain
Keywords: Virtual reality
MeSH Terms: conditions — Gastrointestinal Diseases; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR Arm (Other): Viritual Reality therapy arm. All patients will receive virtual reality therapy.
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Virtual Reality therapy

SUMMARY:
The purpose of this study is to determine if virtual reality (VR) will improve symptoms in non-cardiac chest pain (NCCP).

DETAILED DESCRIPTION:
The primary aim of this study is to assess the overall feasibility of virtual reality for the treatment of noncardiac chest pain and identify problems, issues, or challenges that may impact the performance of a future clinical trial. As such, the study will focus on willingness to participate, patient adherence, patient retention, and burdensomeness of the intervention and survey instruments. As a lesser objective, we will assess the effectiveness of virtual reality in patients with noncardiac chest pain at improving pain severity, symptom hypervigilance, anxiety, quality of life, and resilience.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of non-cardiac chest pain (recurrent anginal-like or atypical chest pain)
* Negative prior cardiac evaluation (at a minimum, including electrocardiogram)
* Prior esophagogastroduodenoscopy and/or barium esophagram to rule out severe esophagitis, stricture, or motility abnormality

Exclusion Criteria:

* Initiation of a proton pump inhibitor (PPI) within 8 weeks
* Major concomitant illness
* Current drug or alcohol use that that would interfere with adherence to study requirements
* Symptoms of vertigo or dizziness that would limit tolerability of the VR headset

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure changes in GERD symptoms using the GERDQ questionnare | Week 2
  Gastroesophageal reflux disease (GERD) questionnaire (GerdQ) is a 6-item questionnaire (scale from 0 to 18) that measures heartburn, regurgitation, abdominal pain, nausea, sleep disorders, and the over-the-counter (OTC) drugs use. The score predicts the likelihood of GERD, with a score between 11-18 suggesting 89% or greater likelihood.
Measure changes in GERD quality of life using the GERD-HRQL questionnaire | Week 2
  GERD-HRQL- Gastroesophageal reflux disease (GERD) - Health Related Quality of Life (HRQL) The scale has 15 items, which focus on heartburn symptoms, dysphagia, medication effects and health condition. Each item is scored from 0 to 5 (maximum score 75), with a higher score indicating a better QOL
Measure changes in esophageal symptom specific anxiety using the EHAS questionnaire | Week 2
  The esophageal hypervigilance and anxiety scale (EHAS) The EHAS is a 15-item measure with two factors evaluating esophageal hypervigilance and symptom specific anxiety scored on a 0-4 Likert scale. Items are summed to yield a total score ranging from 0 - 60 (Greater hypervigilance/anxiety).
Measure changes in GI symptom severity using the PAGI-SYM questionnaire | Week 2
  Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) The PAGI-SYM includes 6 subscales ranging from 0 (none) to 5 (very severe): heartburn/regurgitation, fullness/early satiety, nausea/vomiting, bloating, upper abdominal pain, and lower abdominal pain.
Measure changes in GI related patient assessment of quality of life using PAGI-QOL | Week 2
  Patient Assessment of Gastrointestinal Disorders-Quality of Life (PAGI-QOL) The PAGI-QOL Is an instrument scoring 30 factors each from 0 (none of the time) to 5 (all of the time). Symptoms are assessed over a 2 week period and include the 5 domains daily activities, clothing, diet and food habits, psychological well-being/distress, and relationships.

SECONDARY OUTCOMES:
Measure changes in anxiety and depression using the HADs scale | Week 2
  The Hospital Anxiety and Depression Scale (HADs) consists of 14 items and consists of two subscales: anxiety and depression. Each item is rated on a four-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represents 'borderline' and 0-7 'normal'.
Measure changes in resilience using the brief resilience scale | Week 2
  The brief resilience scale is a 6 question survey assessing resiliency with questions assessed by a 5 point Likert scale.
  12-item short form survey (SF-12). The SF-12 is a 12 question survey assessing the impact of health on a patient's everyday life. The questions assess 8 domains including physical activities, social activities, pain, mental health, vitality, general health perceptions and limitations related to physical and emotional problems.

CONTACTS AND LOCATIONS:
Overall Officials: Andree Koop, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials